CLINICAL TRIAL: NCT02269657
Title: Patients' Arm Positioning in the EOS® Stereoradiography System: Study the Sagittal Spinal Parameters and Postural Balance in EOS® Full Spine X-rays in Scoliosis
Brief Title: Adolescent Idiopathic Scoliosis (AIS) Patient Positioning in EOS System®
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: EOS imaging Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-011016
Record Dates: First submitted 2014-10-13; First posted 2014-10-21 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Postural balance; Lordosis; Kyphosis; X-rays
MeSH Terms: conditions — Scoliosis; Lordosis; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subject Cohort: Two bi-planar full spinal X-rays will be taken using the EOS® imaging system with subjects standing in two different positions. The first x-ray will be taken while the subject's hands and forearms in front of them on the wall vertically. A second image will be taken while the subject's knuckles loosely placed on ipsi-lateral clavicles. A pressure mat will record the magnitude of pressure under the subjects' feet during each set of images. A third set of pressure mat recordings will be obtained while the subject is in a natural standing position with both arms hanging on either side (no x-ray images will be taking in this position).
  Interventions: Device: EOS® imaging system

INTERVENTIONS:
Device: EOS® imaging system — The EOS® imaging system is a low dose, 3-dimensional imaging system that provides weight bearing images which provide visual information with respect to the interaction between the joints and the rest of the musculoskeletal system, particularly the spine, hips and legs. The imaging system is used for clinical purposes with additional images captured as part of this study to collect data from subjects in two different arm positions during imaging.

SUMMARY:
The EOS® imaging system, a new imaging modality which offers low dose, weight bearing and full body X-ray imaging, requires a new standing position where patients put their hands and forearms on the wall vertically for stability. Although this method provides enough support for the patients during the extended X-ray acquisition time, its impact on the postural balance and sagittal profile of the spine and sacro-pelvic parameters has not been evaluated. The goal of this study is to identify the impact of patients' arm positioning on the sagittal profile and postural balance of the patient and subsequently propose a standardized method for full spine X-ray acquisition in the EOS® imaging system.

DETAILED DESCRIPTION:
Spino-pelvic sagittal analysis and postural assessment are important parameters in adolescent idiopathic scoliosis (AIS) treatment and surgical planning.The three-dimensional (3D) shape of the spine is impacted by the patients' posture particularly in adolescents with flexible spinal curves. The latter highlights the importance of the patients' positioning during X-ray acquisition in order to avoid any misleading measurements that may adversely impact monitoring and surgical curve correction in AIS.

Participating subjects will undergo two bi-planar X-rays in different positions. The positions will be instructed by the means of graphical presentation and verbal explanation by the radiology technician. The first standing position in the EOS® imaging system for full spinal X-ray acquisition will consist of putting both hands and forearms in front of the subject on the wall vertically. In the second position, knuckles are loosely placed on ipsi-lateral clavicles. Bi-planar X-rays will be taken in the EOS® imaging system for both positions.

Moreover to compare the postural balance of the patient in the two described positions, a pressure mat will be placed in the EOS® system. The pressure mat will be calibrated with the EOS® system and permits to identify the position of the center of pressure (COP) with respect to the anatomical landmarks. The magnitude of pressure under the patients' feet will be measured during each X-ray and compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 10-18
* Diagnosis of adolescent idiopathic scoliosis
* Prescribed bi-planar full spine X-ray images
* Must be able to stand still for 10 seconds without any support
* Must be able to follow verbal and visual instruction

Exclusion Criteria:

* Previous surgical treatment
* Diagnosis of a neuro-muscular disorder
* Have supernumerary vertebrae, congenital deformities, spondylolisthesis, or spina bifida
* Have any other musculoskeletal disorder that impacts standing balance such as hip, knee, ankle pain and instability or lower back pain
* BMI higher than 30
* Pregnant or lactating females
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Outpatient adolescent idiopathic scoliosis patients visiting the orthopedic clinic at Children's Hospital of Philadelphia who require bi-plannar full spine x-ray imaging for clinical purposes.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saba Pasha, PhD, Principal Investigator — Children's Surgical Associates
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiable pressure mat data from select subjects that is recorded during this study will be shared with investigators at this institution working on another approved study which requires pre-surgical pressure mat data. Many subjects in the companion study will have already undergone surgery, yet none in the current study will have at the time pressure mat data is recorded. Thus this data will be shared. Data will be stored in a password protected file on a secure shared drive and is only accessible by IRB-approved members of the current and companion study teams.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient adolescent idiopathic scoliosis (AIS) patients were prospectively recruited from the orthopedic clinic at Children's Hospital of Philadelphia. Males and females ages 10-18 years with a diagnosis of AIS with no previous spinal surgery were included.
Groups:
- Subject Cohort: Two bi-planar full spinal X-ray were taken using the EOS® imaging system with subjects standing in two different positions. The first x-ray was taken while the subject's hands and forearms in front of them on the wall vertically. A second image was taken while the subject's knuckles loosely placed on ipsi-lateral clavicles. A pressure mat recorded the magnitude of pressure under the subjects' feet during each set of images.
Period: Overall Study
Arm/Group | Subject Cohort
Started | 40
Completed | 37
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: 40 subjects consented to participate; however 3 were subsequently deemed ineligible. The analysis population only includes the 37 eligible subjects.
Groups:
- Subject Cohort: Two bi-planar full spinal X-rays were taken using the EOS® imaging system with subjects standing in two different positions. The first x-ray was taken while the subject's hands and forearms in front of them on the wall vertically. A second image was taken while the subject's knuckles loosely placed on ipsi-lateral clavicles. A pressure mat recorded the magnitude of pressure under the subjects' feet during each set of images.
Arm/Group | Subject Cohort
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.7)
Gender [Count of Participants; unit: Participants]
  Female | 30
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Impact of the Patients' Arm Positioning on Clinical Evaluation of Bi-planar Spinal X-rays Using the EOS System - Spinal Sagittal Plane Parameters
Description: Spinal (coronal and sagittal) and sacro-pelvic parameters were used to evaluate the equivalence between the spinal and pelvic parameters in the two arm positions.
Time Frame: Up to 30 minutes
Population: Each enrolled subject completed bi-planar full spinal x-rays in each of the two positions.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Wall Position: Subjects stood with a 90 degree shoulder and elbow flexion with forearms and palms on the wall in front of them. Bi-planar low dose x-ray images of the spine and pelvis were taken with a pressure mat recording the position of the arm center of pressure in each arm position. Spinal and pelvic parameters and standing balance in different arm positions were measured.
- Clavicle Position: Subjects stood with a 45 degree shoulder flexion with their knuckles on their clavicles. Bi-planar low dose x-ray images of the spine and pelvis were taken with a pressure mat recording the position of the arm center of pressure in each arm position. Spinal and pelvic parameters and standing balance in different arm positions were measured.
Arm/Group | Wall Position | Clavicle Position
Number analyzed (Participants) | 37 | 37
degrees
  Cervical lordosis | 5.9 (25.4) | 7.6 (24.9)
  T1-T12 Thoracic kyphosis | 29.5 (10.3) | 33.55 (12.5)
  T4-T12 Thoracic kyphosis | 19.8 (10.4) | 22.6 (10.6)
  L1-L5 Lumbar lordosis | 46.1 (13.9) | 45.5 (13.1)
  L1-S1 Lumbar lordosis | 56.3 (13.7) | 57.7 (13.1)

2. Primary Outcome: Impact of the Patients' Arm Positioning on Clinical Evaluation of Bi-planar Spinal X-rays Using the EOS System - Frontal Spinal Plane Parameters
Description: as for outcome 1
Time Frame: Up to 30 minutes
Population: Each enrolled subject completed bi-planar full spinal x-rays in each of the two positions.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Wall Position | Clavicle Position
Number analyzed (Participants) | 37 | 37
degrees
  Proximal thoracic Cobb | 23.5 (12.6) | 27.7 (7.8)
  Main thoracic Cobb | 50.3 (17.5) | 51.3 (17.2)
  Lumbar Cobb | 43.9 (16.4) | 41.3 (17.7)
  T1 tilt | -4.1 (8.8) | -8.6 (11.3)
  L4 tilt | -8.2 (12.5) | -5.3 (9.3)
  Main thoracic apical vertibral translation | -3.4 (2.4) | -2.3 (3.2)
  Lumbar apical vertebral translation | 1.9 (2.3) | 1.0 (2.4)

3. Primary Outcome: Impact of the Patients' Arm Positioning on Clinical Evaluation of Bi-planar Spinal X-rays Using the EOS System - Transverse Plane Parameters
Description: as for outcome 1
Time Frame: Up to 30 minutes
Population: Each enrolled subject completed bi-planar full spinal x-rays in each of the two positions.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Wall Position | Clavicle Position
Number analyzed (Participants) | 37 | 37
degrees
  Main thoracic apical vertebral rotation | -10.8 (16.5) | -12.0 (9.8)
  Lumbar apical vertebral rotation | 14.6 (9.9) | 13.7 (8.8)

4. Primary Outcome: Impact of the Patients' Arm Positioning on Clinical Evaluation of Bi-planar Spinal X-rays Using the EOS System - Pelvic Sagittal Plane Parameters
Description: as for outcome 1
Time Frame: Up to 30 minutes
Population: Each enrolled subject completed bi-planar full spinal x-rays in each of the two positions.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Wall Position | Clavicle Position
Number analyzed (Participants) | 37 | 37
degrees
  Pelvic incidence | 51.0 (14.8) | 50.6 (14.3)
  Sacral slope | 44.1 (12.4) | 49.9 (15.6)
  Pelvic tilt | 6.8 (8.8) | 9.5 (11.2)
  Anterior pelvic plane inclination | 5.4 (8.1) | 4.1 (6.9)

5. Primary Outcome: Impact of the Patients' Arm Positioning on Clinical Evaluation of Bi-planar Spinal X-rays Using the EOS System - Pressure Mat Parameters
Description: Spinal (coronal and sagittal) and sacro-pelvic parameters were used to evaluate the equivalence between the spinal and pelvic parameters in the two arm positions. Images were only recorded during the wall and clavicle position, not during the natural standing position. Pressure mat parameters were recorded for both arm positions and compared to the natural standing position (arms hanging on either side).
Time Frame: Up to 30 minutes
Population: Each enrolled subject completed bi-planar full spinal x-rays in each of the two positions and pressure mat recording in the two positions and the natural standing position.
Measure: Mean (Standard Deviation); unit: percentage of pressure under
Groups:
- Natural Standing Position: Subjects stood with their arms hanging on either side. Images were not taken but a pressure mat recording of the position of the arm center of pressure during this arm position was recorded.
Arm/Group | Wall Position | Clavicle Position | Natural Standing Position
Number analyzed (Participants) | 37 | 37 | 37
percentage of pressure under
  Right foot | 44.9 (4.5) | 44.0 (5.6) | 44.2 (6.2)
  Left foot | 55.0 (4.5) | 55.9 (5.6) | 55.7 (6.1)
  Front of right foot | 34.2 (7.1) | 40.1 (10.4) | 41.6 (8.6)
  Back of right foot | 65.7 (7.1) | 59.8 (10.4) | 58.4 (8.7)
  Front of left foot | 35.7 (9.2) | 39.3 (9.5) | 41.6 (9.8)
  Back of left foot | 64.2 (9.2) | 60.6 (9.5) | 58.3 (9.8)

ADVERSE EVENTS:
Time Frame: 30 Minutes
Arm/Group | Subject Cohort
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes